CLINICAL TRIAL: NCT07039643
Title: The Pilates Method in the Rehabilitation of Achilles Tendinopathy - A Randomised Controlled Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, AIKATERINI SIVRIKA, PT, MSc, PhD(c), Physiotherapy Department of the University of West Attica, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 41860/07-05-2025
Record Dates: First submitted 2025-06-17; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Achilles Tendinopathy; Achilles Tendinopathy (AT); Eccentric Exercise; Pilates Method; Pilates Exercise
Keywords: Achilles tendinopathy; Achilles Tendon injuries; exercise; Rehabilitation; Pilates exercise; Pilates method; Pilates
MeSH Terms: conditions — Motor Activity | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: Parallel Assignment. This is a randomised controlled trial with primary end point at 8 weeks for the intervention group and second primary point at 12 weeks while the end point for the control group will be at 12 weeks. Participants will be allocated randomly into two groups (intervention and control).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Pilates Group (Experimental): Group A will follow exercise sessions based on the Pilates method. The protocol will be determined and performed twice a week for 60 seconds, for 8 weeks with a 12 week follow-up. The Pilates will be performed on Reformer equipment and at the final stages jumboard will be added.
  Interventions: Other: Pilates exercise
- Group B: Alfredson Group (Active Comparator): Group B will follow the Alfredson Protocol at home with a diary. Instructions at the beginning will ensure the correct execution while there will be communication once a week to ensure the commitment and compliance. Participants will have to perform 3 sets of 15 repetitions of each exercise 7 days a week for 12 weeks.
  Interventions: Other: Alfredson protocol

INTERVENTIONS:
Other: Pilates exercise — This study investigates a novel Pilates-based rehabilitation program for Achilles tendinopathy (AT). While eccentric loading is the standard treatment, many patients experience persistent symptoms or poor adherence. Pilates emphasizes core stability, neuromuscular control, and functional movement, offering a holistic approach that addresses kinetic chain dysfunction and movement impairments often overlooked in standard protocols. This trial will assess the feasibility and effectiveness of Pilates in improving pain, function, and movement quality in adults with AT. To our knowledge, this is the first clinical trial to evaluate Pilates as a targeted intervention for AT.
  Arms: Group A: Pilates Group
Other: Alfredson protocol — At our knowledge this is the first study that will compare the most popular protocol in Achilles Tendinopathy to an alternative exercise method
  Arms: Group B: Alfredson Group

SUMMARY:
Achilles Tendinopathy (AT) is characterized by pain, swelling and dysfunction. Rehabilitation strategies focus on conservative treatment, with eccentric exercise being the main and most popular option. Patient education based on the biopsychosocial model is considered important for effective self-management, including modification of activities and loads and pain monitoring. Established exercise protocols are applied in rehabilitation, with eccentric, eccentric- concentric combinations and high-resistance exercises performed at a slow pace being the most popular. The Pilates method , which has gained popularity in recent years, focuses on core stabilization, motor control, correct posture through respiratory patterns during execution as well as flow and mindfulness and is applied to the rehabilitation of various musculoskeletal disorders. Although there is a research background in rehabilitation, the data for its application in AT are limited. The present study aims to investigate the integration of Pilates into clinical practice for AT.

DETAILED DESCRIPTION:
Achilles Tendinopathy (AT) is a common condition characterized by pain, swelling, and functional impairment. This condition often occurs after overuse activities and is common in athletes involved in both recreational and professional sports, especially runners, as well as in the general population. Within the context of sports activities and in addition to sports, certain risk factors have been identified that increase the prevalence. In general, these factors include age, gender, biomechanical factors, changes in training plan, inappropriate footwear, hard training surfaces and others. The lifetime prevalence of AT has been estimated at 6% in the general population, aged 18-65 years. In children and adolescents (<18 years), the prevalence ranges from 8% to 33% and is higher in boys. In the general population of runners and marathon athletes, the reported prevalence of Achilles Tendinopathy ranges from 6.2% - 9.5% and 2.0% - 18.5% respectively, while other studies in runners have reported lifetime prevalence reaching 36% for shorter distance runners and 52% for middle and long distance runners. In runners, the risk has been estimated to be 10 times greater than in the general population.

Studies have also examined the prevalence of AT among different types of the disorder. The prevalence of insertional AT has been reported to be approximately 4% in the general population and 14% in the athletic population, with quite high prevalence rates of up to 21% in runners. Regarding mid-portion AT, the incidence rate was estimated at 1.85 per 1,000 registered medical patients in the Dutch health system, in a cohort study including 57,725 individuals. In the adult population, aged 21-60 years, the incidence rate was 2.35 per 1,000 individuals, while in 35% of cases a relationship to sports activity was recorded. In addition to the high incidence, there is a significant negative impact of AT on quality of life, work productivity and overall healthcare costs. A recent study estimated that this amounts to approximately €840 per patient, for those undergoing conservative treatment per year.

A significant proportion of patients with AT develop chronic symptoms lasting up to 10 years. A ten-year follow-up study investigated the chronicity of symptoms in a sample of 43 patients with mid-portion AT and found that 19% of those who had received conservative treatment still had symptoms after 10 years, while only 1/3 were able to perform sports activities without pain at the level before the onset of AT. The chronicity of symptoms seems to contribute to large variations in recovery rates.

In the literature and clinical practice, a wide range of treatment methods for Achilles tendonitis are described and applied with varying levels of effectiveness. Patient education through the lens of the biopsychosocial model is particularly important throughout the rehabilitation period by developing conditions of trust-compliance in self-management which includes modification of applied loads and implementation of exercise strategies as exercise programs play a decisive role in AT. The patient needs a thorough understanding of the purpose of the exercises, the use of the pain monitoring model and the expected prognosis. In general, healthcare providers should provide the patient with advice and knowledge about the condition, prognosis and pain, always taking into account the psychological factors that may have an impact. Important points for discussion and advice are the temporary cessation of (sports) activities that cause pain, the gradual increase in the load of (sports) activities and the use of a pain scale to monitor pain levels.

Exercise is currently the cornerstone in the rehabilitation of AT, as it has been shown to contribute significantly to improving functionality and reducing pain. Mechanical loading on the tendon is crucial to keeping it healthy and strong. Animal studies provide evidence that the tendon is positively affected by physical exercise as it becomes larger, stronger, and more resistant to injury. Exercise has also been shown to increase blood circulation and enhance collagen synthesis in the Achilles tendon.

Despite the different approaches that have been proposed in the literature, eccentric exercise remains the most widely used first-line treatment today, as shown by studies conducted in samples of physiotherapists in various countries. Research found the use of many types of resistance exercises for the management of AT, including isometric, eccentric, concentric and plyometric exercises. Yet, the the majority of programs support eccentric exercise namely the Alfredson protocol. The Alfredson protocol remains the most popular.

A recent systematic review that exclusively examined the application of exercise as a means of rehabilitation for patients with both insertional and mid-portion AT reached the same results. In this study, it was observed that although the combination of concentric-eccentric and high-resistance exercises performed at a slow pace showed positive results, due to the small number of studies and other methodological limitations, eccentric seemed to be more effective.

However, eccentric exercise programs are particularly demanding as the traditional protocol involves completing six sets of exercises, each consisting of 15 repetitions, twice a day for 12 weeks, although later studies showed that a smaller number of repetitions can lead to equivalent positive results. The Alfredson protocol, according to systematic reviews published in recent years, is presented as the most effective in the athletic population, while it is shown to be less effective in the general population and in the elderly. Studies suggest a more personalized exercise program rather than implementing specific protocols with the aim of improving tissue functional capacity through load application and management. In this context, alternative exercise approaches that are widely popular among the population could be implemented in rehabilitation and can have research interest.

Pilates is a popular exercise method that focuses on breathing, central stabilisation, flexibility, motor control, posture, flow and mindfulness. These special characteristics make it suitable for rehabilitation environments, mainly in chronic musculoskeletal disorders. Research on the Pilates method as a means of rehabilitation in musculoskeletal disorders focuses on spinal diseases, while there is research interest in applying the method to the rehabilitation of injuries of the upper and lower extremities. During the last decade, there has been research interest in the rehabilitation of tendinopathies in an effort to create implementation protocols for the part of the population that has difficulty following and executing established protocols.

However, the extent of use of therapeutic Pilates in clinical practice remains unknown, both in the Greek and international contexts, and existing reports are isolated. The lack of data on the application of Pilates in clinical practice limits its further use in rehabilitation in other disorders such as Achilles Tendinopathy, due to the absence of data on the most appropriate programs and their dosage.

The purpose of the present study is to investigate the application of rehabilitation programs for Achilles Tendinopathy, based on the Pilates method, in daily clinical practice. Through this investigation, the aim is to improve the therapeutic effectiveness and promote the integration of the Pilates method in more clinical uses.

Methodology The study will be randomized. The groups will be randomly assigned and will be equivalent (each patient will have the same chance of being assigned to either group) and double-blind (the patients will not know which protocol is being applied).

Patients will be approached through other healthcare professionals and referred to the principal investigator.

The principal investigator will be responsible for the delivery and collection of the completed information-consent form which will be completed by the prospective patients at the site where the study will be conducted, at Physioway physiotherapy center . At this stage, pseudonymization will be carried out by the principal investigator in order to ensure the protection of the patients' personal data. Subsequently, the person responsible for sampling, who will not participate in any of the subsequent stages of the study, will interview each patient individually to verify basic demographic, somatometric and clinical characteristics and their suitability for participation in the study based on specific acceptance and exclusion criteria according to their history and clinical assessment:

* Name
* Age
* Sex
* Level from education
* Start and duration of symptoms
* Previous treatments The data collected during the assessments will be, as previously mentioned, pseudonymized with a code number for the purpose of protecting personal data as well as for blinding purposes. Only the responsible physiotherapist will have access to the participants' contact details. The research manager who will make the measurements will not know which group each patient has been placed in.

The physiotherapists participating in the study will supervise the participants to ensure the correct execution of the protocols but will not participate in any of the subsequent stages of the study.

The research manager will carry out the measurements and analyze the data with the help of the statistician, a member of the three-member committee . Lamnisos Dimitris.

The paper data will be kept by the principal investigator in a locked drawer in an office with exclusive access by her. The data in electronic form will be kept by the principal investigator on a computer and a file with access codes. The computer has an updated antivirus system. The data will be transmitted in pseudonymized form to the other researchers in order to process, analyze and extract the results. The data will be destroyed after the completion of the collection and processing of the data and specifically by 30/12/25.

Patients will be informed about the content and objectives of the study, as well as their ability to withdraw at any time. They will be required to sign a relevant consent form for participation in the study. At the same time, they will be informed about their ability to file a complaint or grievance. For any grievance regarding the conduct of the research, they can contact the Research Ethics and Conduct Committee of the University of West Attica ( ethics @ uniwa . gr ). For any complaints regarding the management of personal data, they can also contact the Data Protection Officer of the University of West Attica. In case of failure to resolve a potential problem, participants can contact the Data Protection Authority by completing the relevant form found on its website ( complaints@dpa.gr ).

Population Inclusion criteria: Men and women within the age range of 18-40 years with diagnosed tendinopathy will participate in the study. The sample will come from athletes (amateurs and professionals) as the main outcome measure for which the validity and reliability were studied was found to be applicable to this specific population group. Epidemiology, as mentioned above, reports high levels of prevalence of the condition in this population group of athletes. A total of 38-40 patients aged 18-40, residents of Athens, who speak Greek and have been referred by their doctor, physiotherapist or have voluntarily come to the AT with pain will participate in this study. Patients will come after a public invitation for voluntary participation that will be posted on the Panhellenic Association of Physiotherapy page, as well as on all electronic media available to the Association ( Viber , Facebook ). Also, the Hellenic Society of Orthopaedic Surgery and Traumatology (H.E.X.O.T.) and the Hellenic Society of Physical Medicine and Rehabilitation (H.E.F.I.A.) will be asked to host on their pages an invitation for patient referral and participation in the study.

The sample selected to participate in the research will be divided into 2 groups by drawing lots by the responsible professor. The patients will be evaluated and receive treatment at Physioway Physiotherapy Laboratory.

Exclusion criteria: Individuals with a history of surgery on the Achilles tendon and a history of surgery around the ankle will be excluded from the study . Individuals with a history of cancer, other pathological factors and medication that may affect the progression of the condition, chronic cortisone use, as well as individuals who received other conservative treatment in the previous four weeks from their entry into the study will also be excluded.

Research protocol Three physiotherapists with experience in the Pilates method for at least 2 years will participate in the study. These physiotherapists will supervise the correct execution of the protocols but will not participate in any of the subsequent stages of the study.

To determine the required sample size, a power analysis was performed using G * Power software . The analysis was based on the study design ( Repeated Measures ANOVA , mixed model , two groups and three or four measurements) with a significance level (α) of 0.05 and a desired power of 80% (0.80). The effect size ( effect size ) was set at the medium level (0.25), according to the data of the existing literature on corresponding clinical trials. According to the results of the analysis, a total sample of 34 participants (17 people per group) is required for the sufficient statistical power of the study. Taking into account the probability of losses due to dropouts at a rate of 10-15%, it is proposed that the initial sample size be 38-40 people.

The sample will be randomly assigned to two groups that will receive a different intervention. One group (intervention group) will perform exercises based on the Pilates method (based on the results collected from the questionnaire and scoping review )( Sivrika and al ., 2024) and the other group (control group) the Alfredson protocol based on the results of the systematic review ( Sivrika and al ., 2023). The content of each session will consist of warm-up exercises, exercises according to the group to which each participant belongs and cool-down exercises at the end of each session. The exercises will be modified-evolved depending on the stage in which each participant is.

The frequency of the intervention will be 8 weeks with a follow-up at 12 weeks for the intervention group and 12 weeks for the control group.

The intervention group will follow a Pilates program for 8 weeks with a frequency of 2 times a week. The duration of each session will be 60 minutes and the number of repetitions in each applied exercise will be 10 repetitions (results from scoping review ). The exercise program will be based on the results of the questionnaire in the community of Physical Therapists and the basic principles of the method.

The control group will perform the Alfredson protocol , which will include exercises with the knee extended and bent. Patients will perform the protocol on their own following instructions and a performance diary that they will receive from one of the Physical Therapists of the research team. The specific Physical Therapist will also undertake communication once a week with the patients in order to ensure compliance and correct performance. The protocol will include performing three sets of 15 repetitions twice a day. The load will be determined by the stage and symptoms of each patient. Patients will be instructed during the weeks to continue activities such as walking or running only if their symptoms do not increase by 4-5 points on the pain scale.

Control Group Protocol Purpose : The control group will follow an eccentric exercise program based on the Alfredson protocol ( Alfredson and al ., 1998), modified to adapt to the individual needs of the participants.

Program Duration : 12 weeks. Frequency : 2 times a day

Program Structure :

The first stage will involve preparing patients for inclusion in the study and learning proper technique. Emphasis will be placed on the precise execution of the exercises to maximize benefit and avoid injury.

Patients will be given an exercise diary for compliance purposes and instructed to complete the diary daily.

The exercise program will include the basic exercise , i.e. applying eccentric load to the Achilles tendon with the knee in extension and flexion. The exercise will be performed with the affected leg. Participants will step up using both legs and slowly (3 seconds) step down with the affected leg. Participants will perform 3 sets of 15 repetitions for each exercise 7 days a week for 12 weeks. A progressive increase in load based on pain (use of a weight bag) will be applied when there is no pain or the pain level is tolerable and does not exceed 4-5 units on the VAS scale . Patients will be instructed to continue activities such as walking or light running only in case there is no increase in symptoms or impairment of functional capacity. They will also be advised, if there is no increase in pain or dysfunction during the study, to begin gentle walking or light running on a flat surface for a short period of time until the completion of the study in order to conduct the results and to prevent any possible recurrence of symptoms or dysfunction that would affect the outcome of the study.

Intervention Team Protocol Purpose : The intervention team will perform exercises based on the Pilates method with the help of Reformer equipment . The dosage will be determined based on the findings of the scoping review, while the results of the questionnaire will be used to formulate the protocol, adapted to the needs of the participants.

Program Duration : 8 weeks. Frequency of Sessions : 2 times a week. Session Duration : 60 minutes per session.

Program structure:

In the first stage, the basic principles of the method will be learned. The implementation of Pilates exercises will be carried out with the help of the Reformer , while in the final stages, the Jumboard platform will be used .

The program includes exercises on the footbar with both feet in all positions. In the position where the feet are in plantar flexion, the exercise will be performed and alternately. Then the bridges will be performed ( bottom lift and bottom lift with extension). The exercise program will continue with isometric exercises on both legs for 45 seconds using high resistance with the knee in extension and flexion (bridge position on the bed). The repetitions will be 10 in total. Isometrics of 30 seconds single-leg on the affected leg, 10 repetitions with the knee in extension and flexion.

Then, with the healthy leg on the footbar , concentric loading and eccentric loading will be performed with both legs. Then concentric with the healthy leg and return with the affected leg (eccentric). Progressively, the concentric -eccentric exercise is performed with the affected leg and less resistance. The same exercise is performed with the pelvis in a bridge position at the beginning with both legs and progressively with the affected leg with less resistance. Progressively, the jumpboard platform is placed and at the beginning, the exercise is performed on soft ball on the affected leg, while then bounces are applied initially with both legs, then alternately and in the final stage with the affected leg. In the last stage, the landing is performed with the affected leg in plantar flexion.

In the same position, lower limb stretching exercises will be performed with the help of straps ( e.g. adductors & hamstrings stretch ). In a standing position, the exercises skating , side splits , as well as up & down exercises stretches , shoulder push and hamstring curl to enhance core stabilization and a holistic approach.

Finally, scooter exercise, with the coordination of the upper limbs which simulates walking and running and standing lunge to enhance the flexibility of lower limb muscles in a functional position.

Outcome Measures

The following outcome measures will be used:

1. TENDINS - A questionnaire TENDINS - A is a new, valid and reliable outcome measure that assesses pain, symptoms and physical activity. It exhibits adequate content validity and is considered the most representative tool for quantifying the effectiveness of interventions in Achilles tendon rehabilitation ( Murphy and al ., 2024). The study on cross-cultural adaptation-translation and validity-reliability in the Greek language received approval from the Hellenic National Institute of Language and Culture with protocol number 102962/05-11-2024 . The results of the study were used to determine the characteristics of the main study sample.
2. Single heel rise test ) The heel rise test records the number of repetitions until pain or fatigue occurs, while its effectiveness in assessing functional recovery has been documented with the maximum strength of recommendation (A) ( Silbernagel and al ., 2020).
3. Tampa Scale for Kinesiophobia ( TSK) Fear of movement and physical activity will be assessed with the Greek version of the Tampa Scale for Kinesiophobia ( Georgoudis) and al ., 2005; Miller and al ., 1991). The TSK is a valid and reliable self-assessment tool that includes two subscales : activity avoidance and bodily focus-perception.

   The total score ranges from 17 to 68, where 17 indicates no kinesiophobia and 68 indicates severe kinesiophobia . A score > 37 indicates the presence of kinesiophobia .
4. VAS pain scale ( Visual Analogue Scale ) Data collection will take place at 4 time points for both groups 0,4,8,12 weeks.

Statistical analysis Data analysis and statistical processing will be carried out using Microsoft programs. Excel and IBM SPSS Inc. Statistics for Windows , version 29.0.

Normal graphs. Q - Q Plot while the statistician with the Shapiro - Wilk test. Descriptive statistical analysis will be performed on demographic data at baseline and outcome measures at each subsequent time assessment at 3 time points for the control group, 0,6,12 weeks and at 3 time points for the intervention group, 0,4,8 weeks.

Qualitative data will be summarized and presented using frequency tables and graphs. Quantitative data will be summarized and presented using descriptive statistics tables. The mean and standard deviation will be used to summarize the typical value and variability. When there are outliers , the median and interquartile range will be used.

To compare the results between the groups of each therapeutic intervention ( Pilates and control), the t -test for independent samples will be used. For the comparison of repeated measurements in the time factor within each group, a statistical test of sphericity will be performed using the Mauchly criterion and one-way analysis of variance ( one - way ANOVA ) followed by parametric pairwise comparison of samples with Bonferroni correction .

In case the criteria for parametric statistics are not met, non-parametric tests will be applied, Mann - Whitney test for comparing two samples (instead of Independent samples t - test ) and Friedman test for more than two samples (instead of repeated measures one - way ANOVA ).

The level of statistical significance will be set at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women within the age range of 18-40 years with diagnosed Achilles Tendinopathy.
2. Ability to provide consent and good knowledge of the Greek language

Exclusion Criteria:

1. Previous surgery in Achilles Tendon
2. Previous surgery in foot
3. Previous history of cancer, systemic diseases or autoimmune in the acute phase of symptoms
4. Previous use of medication or injections for the AT for the last 4 weeks
5. Previous long-term use of cortisone
6. Participation in a physical or other conservative therapy program for the last 4 weeks

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
TENDINS-A | Data collection will take place at 4 time points 0,4,8,12 weeks.
  TENDINS - A is a new, valid and reliable outcome measure that assesses pain, symptoms and physical activity. It exhibits adequate content validity and is considered the most representative tool for quantifying the effectiveness of interventions in Achilles tendon rehabilitation . tendinopathy ( Murphy and al ., 2024). The study on cross-cultural adaptation-translation and validity-reliability in the Greek language received approval from the Hellenic National Institute of Language and Culture with protocol number 102962/05-11-2024 . The results of the study were used to determine the characteristics of the main study sample.

SECONDARY OUTCOMES:
Single- leg heel -rise test | Data collection will take place at 4 time points 0,4,8,12 weeks.
  The heel rise test records the number of repetitions until pain or fatigue occurs, while its effectiveness in assessing functional recovery has been documented with the maximum strength of recommendation (A) ( Silbernagel and al ., 2020).
Tampa Scale for Kinesiophobia ( TSK) | Data collection will take place at 4 time points 0,4,8,12 weeks.
  Fear of movement and physical activity will be assessed with the Greek version of the Tampa scale. Scale for Kinesiophobia ( Georgoudis) and al ., 2005; Miller and al ., 1991). The TSK is a valid and reliable self-assessment tool that includes two subscales : activity avoidance and bodily focus-perception.
  The total score ranges from 17 to 68, where 17 indicates no kinesiophobia and 68 indicates severe kinesiophobia . A score > 37 indicates the presence of kinesiophobia .
VAS scale | Data collection will take place at 4 time points 0,4,8,12 weeks.
  Visual Analogue Scale for Pain describes pain from 0 to 10. O dercribes a condition free of pain while 10 derscribes most pain.

CONTACTS AND LOCATIONS:
Overall Officials: AIKATERINI P SIVRIKA, PhDc, Principal Investigator — University of West Attica; Dimitrios Stasinopoulos, PhD, Study Director — University of West Attica
Locations (1):
- Physiotherapy Department, University of West Attica, Athens, Aigaleo, Greece

IPD SHARING:
Plan to Share IPD: Yes
Only upon agreement by the authors that there will be no further changes and/ or analysis, results of the study will be published and shared. No patient data will be shared to be compliant with the latest GDPR code.
Supporting Information: Study Protocol, CSR
Time Frame: 6 months after publication date and only upon agreement by the authors that there will be no further changes and/or analysis may data be shared.
Access Criteria: It is to the authors discretion to share study data to other researchers.

REFERENCES:
- [Background] Sivrika AP, Kypraios G, Lamnisos D, Georgoudis G, Stasinopoulos D. Pilates Dosage in Rehabilitation of Patients With Musculoskeletal Conditions: A Scoping Review. Sports Health. 2025 Jul;17(4):824-833. doi: 10.1177/19417381241278263. Epub 2024 Sep 19. PMID 39297289
- [Background] Sivrika AP, Papadamou E, Kypraios G, Lamnisos D, Georgoudis G, Stasinopoulos D. Comparability of the Effectiveness of Different Types of Exercise in the Treatment of Achilles Tendinopathy: A Systematic Review. Healthcare (Basel). 2023 Aug 11;11(16):2268. doi: 10.3390/healthcare11162268. PMID 37628466
- [Background] Murphy MC, Newsham-West R, Cook J, Chimenti RL, de Vos RJ, Maffulli N, Malliaras P, Mkumbuzi N, Purdam C, Vosseller JT, Rio EK. TENDINopathy Severity Assessment - Achilles (TENDINS-A): Development and Content Validity Assessment of a New Patient-Reported Outcome Measure for Achilles Tendinopathy. J Orthop Sports Phys Ther. 2024 Jan;54(1):70-85. doi: 10.2519/jospt.2023.11964. PMID 37615161
- [Background] Merry K, MacPherson M, Vis-Dunbar M, Whittaker JL, Gravare Silbernagel K, Scott A. Identifying characteristics of resistance-based therapeutic exercise interventions for Achilles tendinopathy: A scoping review. Phys Ther Sport. 2023 Sep;63:73-94. doi: 10.1016/j.ptsp.2023.06.002. Epub 2023 Jul 1. PMID 37536026
- [Background] Malliaras P. Physiotherapy management of Achilles tendinopathy. J Physiother. 2022 Oct;68(4):221-237. doi: 10.1016/j.jphys.2022.09.010. Epub 2022 Oct 21. No abstract available. PMID 36274038
- [Background] de Vos RJ, van der Vlist AC, Zwerver J, Meuffels DE, Smithuis F, van Ingen R, van der Giesen F, Visser E, Balemans A, Pols M, Veen N, den Ouden M, Weir A. Dutch multidisciplinary guideline on Achilles tendinopathy. Br J Sports Med. 2021 Oct;55(20):1125-1134. doi: 10.1136/bjsports-2020-103867. Epub 2021 Jun 29. PMID 34187784